CLINICAL TRIAL: NCT04119401
Title: Hemorrhoidal Artery Ligation With Doppler Guidance vs Digital Guidance for Grade II-III Hemorrhoidal Disease Treatment: Randomized Controlled Trial
Brief Title: Hemorrhoid Artery LigatioN Without Doppler Trial
Acronym: HAND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Russian Society of Colorectal Surgeons (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 683473
Record Dates: First submitted 2019-10-06; First posted 2019-10-08 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Hemorrhoids
Keywords: hemorrhoids; hemorrhoidal piles; prolapse; doppler guided ligation; finger-guided artery ligation
MeSH Terms: conditions — Hemorrhoids; Prolapse

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- doppler-guided (Active Comparator): ligation of hemorrhoidal arteries with doppler guidance
  Interventions: Procedure: doppler-guided hemorrhoidal artery ligation
- finger-guided group (Experimental): ligation of hemorrhoidal arteries without doppler guidance but with finger detection
  Interventions: Procedure: Finger-guided hemorrhoidal artery ligation

INTERVENTIONS:
Procedure: doppler-guided hemorrhoidal artery ligation — Ligation: a lubricating gel is applied to the tip of the Transanal Hemorrhoidal Dearterialization device and, with the patient in the lithotomy position, the proctoscope is introduced into the anal canal. The terminal branches of the superior rectal artery are detected by the doppler signal 2-3 cm above the dentate line. The tip of the instrument is gently tilted and the arteries are ligated with a Z-shaped stitch using 2:0 braided polyglycolic acid suture inserted using a special needle-holder through an aperture in the operating proctoscope.
  Mucopexy: after the haemorrhoid artery ligation, the suture is continued with three to five sutures applied 5 mm apart, making sure that the last is at least 5 mm above the dentate line. The suture is then tied to create a hemorrhoidopexy. The procedure is repeated after all detected artery ligations.
  Arms: doppler-guided
Procedure: Finger-guided hemorrhoidal artery ligation — Ligation: the exact placement of all terminal branches of the superior rectal artery are found by intraoperative palpation at anal clock 2-3cm above the anorectal junction. Then arteries are ligated with Z-shaped suture using 2:0 braided polyglycolic suture.
  Mucopexy is then performed in the same technique as in comparative group
  Arms: finger-guided group

SUMMARY:
Hemorrhoidal artery ligation with Doppler guidance (HAL) and suture fixation of hemorrhoidal nodes (RAR) is a popular minimally invasive technique for hemorrhoidal disease (HD) treatment which uses an ultrasound probe to detect hemorrhoidal arteries for further ligation. We hypothesized that ultrasound guidance has no advantages over manual hemorrhoidal arteries detection for HD treatment.

The aim is to compare the results of HAL-RAR procedure in patients with stage II-III HD with Doppler and manual HA detection.

In this ongoing randomized, controlled, single center clinical study 200 patients randomly divided into group A (HAL-RAR with Doppler US navigation) and group B (HAL with manual HA detection and mucopexy) are planned to be included. The primary endpoint was recurrence of any symptoms of HD; secondary endpoints were pain syndrome severity (VAS), treatment satisfaction (1 to 5 points) and need for the drug therapy in 30 days and 8 weeks after surgery.

Ultrasound guidance technology of HAL with mucopexy could have the same efficacy the manual HA detection regarding the HD treatment effectiveness and patient satisfaction.

DETAILED DESCRIPTION:
Hemorrhoidal disease (HD), in its different manifestations, is not only the most frequented grounds of referring for medical attention, but also one of the reasons for the modest deterioration in the quality of life that can possibly result in temporary or permanent reduction of work capacities. Today, the doppler-guided dearterialization of hemorrhoidal arteries and the following suture-fixation mucopexy in the anal canal (synonyms: mucopexy, hemorrhoids lifting, HAL-RAR) is one of the most popular and actively studied methods of the stage II - III hemorrhoidal disease surgical treatment. A number of publications raise an issue whether it is really necessary to use a doppler while the localization of the hemorrhoidal arteries is typical in the vast majority of the observations and can be easily determined on palpation.

The aim of the study is to compare the direct and long-term results of the II - III grade HD surgical treatment with the use of two techniques of the suture ligation of the hemorrhoidal arteries with mucopexy. One of these methods is classic and widely known HAL-RAR, the other one has a principal differ in no-using the doppler to find the arteries, the surgeon defines them on palpation.

The hypothesis of the study is that the digital detection of hemorrhoidal arteries pulsation followed by suture ligation and mucopexy may be no less effective in the treatment of grade II - III hemorrhoids than the use of a doppler guide.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic grade II and III hemorrhoids according to Golligher.
* No other source of anal bleeding than hemorrhoids due to total colonoscopy
* Written voluntary informed consent

Exclusion Criteria:

* Any previous hemorrhoid surgery (including mini invasive procedures)
* Anal fistula
* Chronic anal fissure with severe spasm of anal sphincters
* Any stage colorectal cancer
* Oral anticoagulants for congenital disorders of the coagulation system
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-01-08 (Actual); Primary Completion 2020-10-10 (Estimated); Study Completion 2021-01-11 (Estimated)

PRIMARY OUTCOMES:
recurrence | 2 weeks - 1 year
  The rate of recurrence of any of initial symptoms or appearance of any new symptom of hemorrhoidal disease: anal bleeding during defecation, prolapse of hemorrhoidal piles or both.

SECONDARY OUTCOMES:
Pain score | 2 weeks
  pain score after surgery will be measured by patient-reported pain level using visual scale ranging from 1 to 10 where 1 is "no pain" and 10 - is the the worst pain imaginable.
Patients satisfaction level | 6 month and 1 year
  Patients will be asked to rate their own satisfaction of the procedure on a scale from 1 to 10 (with 10 being the best) and were asked whether the procedure helped their symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Petr Tsarkov, Prof, Principal Investigator — Russian Society of Colorectal Surgeons
Locations (1):
- Clinic of Colorectal and Minimally invasive surgery, Moscow, Russia

REFERENCES:
- [Result] Aigner F, Bodner G, Conrad F, Mbaka G, Kreczy A, Fritsch H. The superior rectal artery and its branching pattern with regard to its clinical influence on ligation techniques for internal hemorrhoids. Am J Surg. 2004 Jan;187(1):102-8. doi: 10.1016/j.amjsurg.2002.11.003. PMID 14706597
- [Result] Brown SR, Tiernan JP, Watson AJM, Biggs K, Shephard N, Wailoo AJ, Bradburn M, Alshreef A, Hind D; HubBLe Study team. Haemorrhoidal artery ligation versus rubber band ligation for the management of symptomatic second-degree and third-degree haemorrhoids (HubBLe): a multicentre, open-label, randomised controlled trial. Lancet. 2016 Jul 23;388(10042):356-364. doi: 10.1016/S0140-6736(16)30584-0. Epub 2016 May 25. PMID 27236344
- [Result] Hoyuela C, Carvajal F, Juvany M, Troyano D, Trias M, Martrat A, Ardid J, Obiols J. HAL-RAR (Doppler guided haemorrhoid artery ligation with recto-anal repair) is a safe and effective procedure for haemorrhoids. Results of a prospective study after two-years follow-up. Int J Surg. 2016 Apr;28:39-44. doi: 10.1016/j.ijsu.2016.02.030. Epub 2016 Feb 10. PMID 26876958
- [Result] Morinaga K, Hasuda K, Ikeda T. A novel therapy for internal hemorrhoids: ligation of the hemorrhoidal artery with a newly devised instrument (Moricorn) in conjunction with a Doppler flowmeter. Am J Gastroenterol. 1995 Apr;90(4):610-3. PMID 7717320
- [Result] Ratto C, Campenni P, Papeo F, Donisi L, Litta F, Parello A. Transanal hemorrhoidal dearterialization (THD) for hemorrhoidal disease: a single-center study on 1000 consecutive cases and a review of the literature. Tech Coloproctol. 2017 Dec;21(12):953-962. doi: 10.1007/s10151-017-1726-5. Epub 2017 Nov 24. PMID 29170839